CLINICAL TRIAL: NCT02026076
Title: Manual Unloading of the Lumbar Spine: Can it Predict Response to Mechanical Traction? A Study or Reliability and Criterion Referenced Predictive Validity
Brief Title: Manual Unloading of the Lumbar Spine: Can it Predict Responders to Mechanical Traction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Andrews University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Manual Unloading
Record Dates: First submitted 2013-11-13; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-11

CONDITIONS: Low Back Pain
Keywords: low back pain; traction; unloading
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- manual unloading (Experimental): All subjects will first undergo a manual unloading test, followed by a single application of mechanical lumbar traction to determine predictive effect
  Interventions: Other: mechanical lumbar traction

INTERVENTIONS:
Other: mechanical lumbar traction — 15 minutes at up to 50% body weight lumbar traction in supine hooklying with split table open

SUMMARY:
This study will seek to determine if 1) the manual unloading test is reliable, and 2)if the immediate response to traction can be determined by using a simple unloading test in standing. The study wil be completed in two parts: 1) a small pilot sample (n=10) to asses both intra and inter tester reliability, and 2) a consecutive sample of 30 patients with low back pain which does not travel below the knee. All subjects will rate their pain on a 100 mm line both at rest and in their most painful direction of movement. A therapist will then unload the patients spine to determine if they feel any relief. All subjects will then undergo a 15 minute bout of intermittent lumbar traction, 30 sec on, 10 sec off at up to 50% body weight. Following traction, all subjects will again rate their pain on a 100 mm line. Subjects will be grouped by response to the initial manual unloading test and assessed for within and between group differences. The study hypothesis is that the manual unloading test is reliable, and that responders to mechanical traction can be accurately identified using a manual unloading test.

DETAILED DESCRIPTION:
This study will consist of two distinct components. Part one will be a reliability study of manual unloading. Two therapists, both familiar with the technique of manual unloading as described by Kaltenborn17, will perform a manual unloading test, blinded to the previous results. Ten consecutive patients will be recruited from a sample of convenience at the University Of Connecticut Health Center Department Of Rehabilitation. This test will be repeated on the same subjects within 7 days of initial testing. Tests of agreement will then be applied to determine intra and inter-rater reliability.

Part two will consist of a trial of lumbar traction in a group of subjects with low back pain without radiculopathy, anticipated n=30. At the time of enrollment, all subjects will complete a standardized informed consent form, detailing all potential risks of the trail. Consent will include permission for demographic data to be obtained from the standard intake form, and kept in a de-identified form in a secure location. All subjects will complete a screening form, which will ensure that the potential subjects do not have any of the excluding factors present. Prior to enrollment, all subjects will complete a standardized medical history form (kept as part of the medical record for all patients), as part of standard departmental practice. Additionally, participants will complete a modified Oswestry questionnaire as well as two 100 mm visual analog scales (VAS), one indicating pain at rest, the other indicating pain in their most provocative test motion (flexion, extension, or side flexion of the lumbar spine). Subjects will then be tested with unloading in standing as described by Kaltenborn. This test involves the therapist applying a low grade lifting force to the patient in a standing position, testing for symptomatic alleviation via the elimination of compression on pain sensitive structures. Results of this test will be coded as (+) relief or (-) relief. Prior to traction application, subjects will undergo a standardized, comprehensive examination (standard of care), which will include screening for exclusion criteria (myotomal weakness, sensation changes, positive neural tension signs). All subjects will be weighed prior to traction application to determine treatment force to be generated. To aid in determining BMI, subjects will also have their height measured. The reference test will consist of a single application of mechanical traction, 15 minutes, 30 seconds on/ 10 seconds off, at 50% of body weight with the treatment table in the opened position, while positioned in a supine, hook lying neutral posture. Post traction, all subjects will repeat AROM measures, and complete a second pair of VAS to determine immediate effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-75
* non-radicular low back pain (LBP)

Exclusion Criteria:

* tumor,
* fracture,
* infectious disorder,
* central nervous system involvement,
* presence of medical red flags,
* absence of LBP,
* radicular leg pain (below the knee),
* pregnancy,
* epidural steroid injection within 4 weeks prior to study involvement,
* previous back surgery,
* workers compensation involvement
* active litigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog pain scale in the most provocative movement | immediate post intervention (within 5 minutes following intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Moss, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States